CLINICAL TRIAL: NCT00283907
Title: Brain Networks Responsible for Sense of Agency: An EEG Study
Brief Title: Brain Networks Responsible for Sense of Agency
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 060084; 06-N-0084
Record Dates: First submitted 2006-01-29; First posted 2006-01-30 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2008-12-16

CONDITIONS: Spatiotemporal Patterns
Keywords: Electroencephalogram (EEG); Sense of Agency; Coherence; Voluntary Movement; Self-Agency; Healthy Volunteer; HV

SUMMARY:
This study of healthy normal volunteers will examine the brain networks involved in people's sense that they control their own movements (sense of agency). Although almost everyone has a sense of agency, some patients (for example, patients with schizophrenia, alien limb phenomena, and others) have movements they think are not under their control. This study will use electroencephalography (EEG) to determine how the normal brain produces the sense of agency. This information will provide a first step in understanding patients with an impaired sense of agency.

Healthy, right-handed men and women 18 years of age and older may be eligible for this study. Candidates are screened with a medical history and neurological examination.

Participants are fitted with a cyberglove device (a lightweight glove with flexible sensors that measure the position and movement of the fingers and wrist) on their right hand. The glove is used to transform the subject's hand and finger motions into real-time digital joint-angle information. Subjects slowly open and close their hand while watching an artificial hand projected on a monitor. They continue practicing the exercise until they are comfortable with the cyberglove and have the sense that the artificial hand is a mirror representation of their own hand, accurately reflecting their hand's movements.

After practicing with the cyberglove, subjects have a functional EEG. For this test, electrodes are placed on the scalp, and brain waves are recorded while the subject opens and closes his or her hand or just watches the computer monitor. The EEG recording takes about 60 minutes.

...

DETAILED DESCRIPTION:
Objective

The purpose of this study is to investigate spatiotemporal patterns of brain networks involved in the sense of agency using high-resolution electroencephalography (EEG).

Study Population

We intend to use 20 right-hand dominant, adult healthy subjects.

Design

The sense of agency (SA) will be modulated using a visual task-based stimulus asking subjects to manipulate the position of an artificial hand projected onto a display. Subjects will use their own right hand to make slow opening/closing movements randomly which will be represented visually with the aid of a Cyberglove. During a behavioral training phase, subjects will practice using the apparatus. The level of control will be randomly changed to one of five states: 100%, 75%, 50%, 25%, 0% control. For secondary analysis, subjects will be asked to report the percentage of control they subjectively feel over the displayed hand. After subjects are comfortable with the apparatus and endorse SA over the displayed hand, they will undergo EEG.

The experimental phase will have five sets of 10 minute recording sessions where the subject is instructed to slowly open and close their hand randomly. The level of control will be changed pseudo-randomly throughout the recording sessions. A control contrast consisting of the subject observing a moving hand will also be integrated into the blocks. An additional control contrast involving the subject moving their hand without visual feedback will also be included. These contrasts will serve in the analysis phase to help eliminate electrophysiological activity related to visual-motor feedback.

A Magnetic Resonance Imaging (MRI) scan of brain will be performed to co-register this EEG data with the anatomical structure. We will integrate physiological (EEG) and anatomical (MRI) data to characterize the regionalization of the task-related brain EEG activity.

Outcome Measures

The primary outcome of this study is the effective connectivity of brain in response to a loss of SA. For this purpose, we will measure the difference of EEG power spectral analysis as well as coherence between 0% and 100 % control. In a secondary analysis, we will investigate the correlation of the EEG measurements with the percent of actual control, and also utilize the individual subject perceptions of percent control during the behavioral training phase as the regressors for activation rather than the objective control settings.

ELIGIBILITY:
* INCLUSION CRITERIA:

Subjects age 18 and older

Subjects must be right-hand dominant (Edinburgh Handedness Quotient greater than 60)

Subjects willing to abstain from caffeine or alcohol for 48 hours prior to the EEG study

EXCLUSION CRITERIA:

Subjects with any abnormal findings on neurological exam

Subjects with any history of brain tumor, stroke, head trauma or a vascular malformation as obtained by history or from imaging studies

Subjects with any history of a severe medical condition, such as cardiovascular disease, which would prevent them from sitting for up to 120 minutes

Subjects without the capacity to give informed consent

Subjects with other restrictions which prevent them from undergoing EEG recordings for up to 60 minutes

Subjects who are taking neuroleptic medications

Subjects are not eligible for Magnetic Resonance Imaging (MRI) scan, if the subjects have pacemakers, intracardiac line, implanted metallic pump, neural stimulator, or a metallic object inside the skull, metal braces, cochlear devices, surgical clips and other metal/magnetic implants; are afraid of being in small spaces; are pregnant

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2006-01-27; Study Completion 2008-12-16

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Gallagher S. Philosophical conceptions of the self: implications for cognitive science. Trends Cogn Sci. 2000 Jan;4(1):14-21. doi: 10.1016/s1364-6613(99)01417-5. PMID 10637618
- [Background] Kircher TT, Leube DT. Self-consciousness, self-agency, and schizophrenia. Conscious Cogn. 2003 Dec;12(4):656-69. doi: 10.1016/s1053-8100(03)00071-0. PMID 14656508
- [Background] Blakemore SJ, Frith CD, Wolpert DM. The cerebellum is involved in predicting the sensory consequences of action. Neuroreport. 2001 Jul 3;12(9):1879-84. doi: 10.1097/00001756-200107030-00023. PMID 11435916